CLINICAL TRIAL: NCT04466579
Title: Influence of Monitoring the Depth of General Anesthesia Upon the Incidence of PONV and Emergence Delirium in Children Undergoing Endoscopic Adenoidectomy in General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-KARIM-14-PONV-ED
Record Dates: First submitted 2020-06-24; First posted 2020-07-10 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Nausea; Postoperative Vomiting; Emergence Delirium
Keywords: postoperative nausea; postoperative vomiting; emergence delirium; bispectral monitor; pediatric anesthesia; adenoidectomy; general anesthesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Emergence Delirium | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study subjects will be randomized into two study arms.
Masking Description: No masking is being used in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIS monitoring (Experimental): Study subjects randomized in this study arm will have the depth of anesthesia controlled with the BIS monitor.
  Interventions: Other: BIS monitor
- Standard care (Active Comparator): Study subjects randomized in this study arm will receive standard anesthesiology care according to the usual procedures used at the study centre.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: BIS monitor — BIS monitor is used to control and monitor the depth of general anesthesia.
  Arms: BIS monitoring
Other: Standard care — Standard anesthesiology care according to the protocol of the study
  Arms: Standard care

SUMMARY:
The study has been designed as a prospective randomized clinical trial. Due to the use of a bispectral (BIS) monitor in the interventional arm, the study will not be blinded for the anesthetist. The total planned number of study subjects is 100. Patients will be randomly randomized upon arrival to the operating theatre (using the envelope method) into the interventional arm (BIS monitoring of the depth of general anesthesia), and into the control group (standard management of general anesthesia to minimum alveolar concentration (MAC) 1,0). The target values of the depth of general anesthesia according to BIS are between 40 and 60.

DETAILED DESCRIPTION:
The condition of postoperative nausea and vomiting (PONV) is defined as nausea and vomiting, which appears within 24 hours after the performance of a surgical/diagnostic procedure in general anesthesia. PONV is perceived as a complication of minor importance in perioperative medicine, nevertheless, it is one of the most frequent causes of morbidity in pediatric patients in the early postoperative period, associated with a number of adverse effects. The incidence of PONV in pediatric age is reported in scientific literature to be between 8.9 and 42 percent. The pathogenesis of PONV is complex and has not been fully clarified yet. The development of PONV depends on individual and anaesthesiology risk factors, and the type of surgical procedure. The use of inhalation anesthetics demonstrably increases the incidence of PONV, especially in the course of the first two hours after the procedure. The need for inhalation anesthetic is individually variable, and it is not possible to empirically define, which dose will lead to an adequate depth of anesthesia. Excessively deep, as well as too shallow anesthesia may result in increasing the incidence of postoperative complications, including PONV. The depth of anesthesia and unconsciousness may be monitored with BIS (bispectral index). The investigators presume that optimization of the supply of inhalation anesthetic according to BIS, so-called BIGA (Bispectral index guided anesthesia) will lead to decreasing the incidence of PONV.

Several clinical studies performed on the adult population have demonstrated that using BIGA leads to a decreased incidence of PONV in adult patients undergoing gynecological procedures. As far as pediatric anesthesiology is concerned, similar studies are still lacking.

Inhalation anesthesia is also associated with another complication in the early postoperative period - so-called emergence delirium (ED). It is a condition of psychomotor restlessness, perception disorders, and excitation of the child observed after completion of anesthesia. The incidence of ED in the pediatric population anesthesia is between 10 and 80 percent, most frequently within the first 10-30 minutes after discontinuation of the administration of anesthetics. The condition is characterized by confusion, loss of orientation, crying, restlessness, and non-cooperation of the child. The causes of ED have not been fully clarified.

One of the possible causes may be the rapid emergence of the child from anesthesia after discontinuation of the inhalation anesthetic. The incidence of ED is highest with Sevoflurane, which is the most frequently used inhalation anesthetic in pediatric anesthesia. Optimization of the depth of general anesthesia and decreasing the consumption of inhalation anesthetic may lead to decreasing the incidence of emergence delirium objectified according to the Paediatric Anaesthesia Emergence Delirium (PAED) score.

The study has been designed as a prospective randomized clinical trial. Due to the use of the BIS monitor in the interventional arm, the study will not be blinded for the anesthetist. The total planned number of study subjects is 100. Patients will be randomly randomized upon arrival to the operating theatre (using the envelope method) into the interventional arm (BIS monitoring of the depth of general anesthesia), and into the control group (standard management of general anesthesia to minimum alveolar concentration (MAC) of 1.0). The target values of the depth of general anesthesia according to BIS are between 40 and 60.

General anesthesia will be administered according to the following uniform anaesthesiology protocol:

Inhalation introduction with Sevoflurane (8% on the vaporizer), in a carrier mixture of gases oxygen : air, with the flow of 41/min and oxygen concentration of 50%. In the intervention group, BIS will be introduced as soon as possible. After achieving a sufficient depth of anesthesia, a peripheral venous catheter will be introduced, followed with intravenous administration of opioid - Sufentanil in the dose of 0.2ucg/kg, and intravenous administration of Paracetamol in the dose of 15mg/kg. The infusion will be administered in the course of the surgical procedure - isotonic crystalloid solution Benelyte in the dose of 10ml/kg/hour. Breathing passageways will be secured with an armed laryngeal mask, according to the standard procedure applied at the author's center. Considering the character of the study, no antiemetic prophylaxis will be administered. After completion of the surgical procedure and emergence from general anesthesia, the child will be transferred to post-anesthesia care unit (PACU), where, apart from the monitoring of vital functions, also the incidence of PONV and the PAED score (in the 10th minute, 30th minute, and 60th minute) will be observed. At the Ear-Nose-Throat (ENT) department, the authors will record the Baxter Retching Faces (BARF) scale in pre-determined time intervals, and the incidence of PONV in the course of the whole hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* 3-8 years of age
* Indication for the performance of endoscopic adenoidectomy in general anesthesia
* ASA I a II
* Consent of a parent/a guardian

Exclusion Criteria:

* ASA III and more
* Disapproval of a parent/a guardian
* Disapproval of the patient
* Allergies to medication used in the course of the study
* Contraindication of inhalation introduction to anesthesia and the way of securing breathing passageways in the study, according to the attending anesthetist

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV | During the hospitalisation of the patient, i.e. up to 5 days
  The incidence of PONV will be observed and recorded using the Baxter Reetching Faces (BARF) scale and recording the number of PONV episodes.
Incidence of ED | During the hospitalisation of the patient, i.e. up to 5 days
  The incidence of ED will be observed and recorded using the PAED score.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Frelich, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
The authors have no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Kovac AL. Management of postoperative nausea and vomiting in children. Paediatr Drugs. 2007;9(1):47-69. doi: 10.2165/00148581-200709010-00005. PMID 17291136
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Dahmani S, Delivet H, Hilly J. Emergence delirium in children: an update. Curr Opin Anaesthesiol. 2014 Jun;27(3):309-15. doi: 10.1097/ACO.0000000000000076. PMID 24784918
- [Background] Locatelli BG, Ingelmo PM, Emre S, Meroni V, Minardi C, Frawley G, Benigni A, Di Marco S, Spotti A, Busi I, Sonzogni V. Emergence delirium in children: a comparison of sevoflurane and desflurane anesthesia using the Paediatric Anesthesia Emergence Delirium scale. Paediatr Anaesth. 2013 Apr;23(4):301-8. doi: 10.1111/pan.12038. Epub 2012 Oct 9. PMID 23043512
- [Derived] Frelich M, Sklienka P, Romanova T, Nemcova S, Bilena M, Strakova H, Lecbychova K, Jor O, Formanek M, Bursa F. The effect of BIS-guided anaesthesia on the incidence of postoperative nausea and vomiting in children: a prospective randomized double-blind study. BMC Anesthesiol. 2024 Jul 9;24(1):228. doi: 10.1186/s12871-024-02610-w. PMID 38982400
- [Derived] Frelich M, Lecbychova K, Vodicka V, Ekrtova T, Sklienka P, Jor O, Strakova H, Bilena M, Formanek M, Bursa F. Effect of BIS-guided anesthesia on emergence delirium following general anesthesia in children: A prospective randomized controlled trial. Anaesth Crit Care Pain Med. 2024 Feb;43(1):101318. doi: 10.1016/j.accpm.2023.101318. Epub 2023 Oct 31. PMID 37918790